CLINICAL TRIAL: NCT01572701
Title: A Phase 1 Pilot Study of 99mTc-MIP-1404 Single Photon Emission Computed Tomography (SPECT)/CT Imaging in Men With Prostate Cancer Undergoing Prostatectomy and/or Pelvic Lymph Node Dissection (PLND)
Brief Title: Pilot Study of 99mTc-MIP-1404 SPECT/CT Imaging in Men With Prostate Cancer Undergoing Prostatectomy and/or Pelvic Lymph Node Dissection
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Molecular Insight Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MIP-TcTx-P104
Record Dates: First submitted 2011-12-05; First posted 2012-04-06 (Estimated); Last update posted 2015-11-25 (Estimated); Status verified 2015-11

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — technetium 99m 1-(1-(2-(bis(carboxymethyl)amino)-2-oxoethyl)-1H-imidazol-2-yl)-2-((1-(2-(bis(carboxymethyl)amino)-2-oxoethyl)-1H-imidazol-2-yl)methyl)-9,14-dioxo-2,8,13,15-tetraazaoctadecane-7,12,16,18-tetracarboxylic acid)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 20 (±3) mCi of study drug (Experimental)
  Interventions: Drug: 99mTc-MIP-1404

INTERVENTIONS:
Drug: 99mTc-MIP-1404 — 20 (±3) mCi of study drug will be administered by IV injection as a slow bolus and flushed with approximately 10 mL of saline

SUMMARY:
This is a single arm, open label study of up to 24 high risk prostate cancer patients scheduled for prostatectomy and/or pelvic lymph node dissection. Patients receive a single IV dose of 99mTc-MIP-1404 (study drug) followed by SPECT/CT scan 3-6 hours after injection. As standard of care, patients will undergo prostatectomy and/or pelvic lymph node dissection (PLND) within two weeks of study drug dosing. Patients may receive a second injection of study drug within 24 hours of surgery to measure activity counts in tissue samples post-surgery, but prior to pathology processing. 99mTc-MIP-1404 image data will be evaluated for visible uptake and compared with histopathology.

ELIGIBILITY:
Inclusion Criteria:

1. Male aged 21 years or older.
2. Ability to provide signed informed consent and willingness to comply with protocol requirements.
3. Past biopsy indicating the presence of adenocarcinoma of the prostate gland.
4. Participant is deemed to be high-risk with potential for pelvic lymph node involvement. The criteria for high-risk are:

   * Patient has PSA value >10 and clinical stage T2 or higher, and Gleason score 8, 9 or 10.
   * Patient has PSA value >20 and clinical stage T2 or higher, and Gleason score
5. Participant is or will be scheduled to undergo standard of care prostatectomy and/or pelvic lymph node dissection.
6. Have had (within previous 2 months) or will undergo diagnostic CT or MRI imaging prior to surgery.
7. Have had (within previous 2 months) or will undergo bone scan imaging prior to surgery.
8. Participants must agree to use an acceptable form of birth control throughout the study period. Participants must use condoms for a period of seven days after each injection, if engaged in sexual activity.

Exclusion Criteria:

1. Participants for whom participating would significantly delay the scheduled standard of care therapy.
2. Participants administered a radioisotope within 5 physical half lives prior to study enrollment.
3. Participants with any medical condition or other circumstances that, in the opinion of the Investigator, would significantly decrease obtaining reliable data, achieving study objectives or completing the study.

Min Age: 21 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2012-01; Primary Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Tissue distribution of 20 (± 3) mCi 99mTc-MIP-1404 | Post-procedure
  99mTc-MIP-1404 image data will be evaluated for visible uptake and compared with histopathology.

SECONDARY OUTCOMES:
Safety of 99mTc-MIP-1404: Change in Vital Signs from Pre-Dose to Post-Dose | Vital signs measurements will be measured, an expected average of 30 minutes before and after study drug injection
  Summary tables will present change from pre-dose to post-dose vital signs measurements.
Intensity of 99mTc-MIP-1404 Uptake with Respect to PSMA expression | Post-procedure
  99mTc-MIP-1404 image data will be evaluated for visible uptake and compared with histopathology.
Safety of 99mTc-MIP-1404: Summary of Treatment-Emergent Adverse Events (TEAEs) | Adverse events will be assessed for the duration of the study participation, an expected average of 3 weeks
  TEAEs will be summarized by the Medical Dictionary for Regulatory Activities (MedDRA) body system and preferred term, by intensity, and by causal relationship to study agent.

CONTACTS AND LOCATIONS:
Overall Officials: Douglas S Scherr, MD, Principal Investigator — New York Presbyterian Hospital - Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College, New York, New York, United States

REFERENCES:
- [Background] Jung JA, Coakley FV, Vigneron DB, Swanson MG, Qayyum A, Weinberg V, Jones KD, Carroll PR, Kurhanewicz J. Prostate depiction at endorectal MR spectroscopic imaging: investigation of a standardized evaluation system. Radiology. 2004 Dec;233(3):701-8. doi: 10.1148/radiol.2333030672. PMID 15564406
- [Background] Swindle P, Eastham JA, Ohori M, Kattan MW, Wheeler T, Maru N, Slawin K, Scardino PT. Do margins matter? The prognostic significance of positive surgical margins in radical prostatectomy specimens. J Urol. 2008 May;179(5 Suppl):S47-51. doi: 10.1016/j.juro.2008.03.137. PMID 18405751
- [Background] Hocht S, Wiegel T, Bottke D, Jentsch H, Sternemann M, Rosenthal P, Hinkelbein W. Computed tomogram prior to prostatectomy. Advantage in defining planning target volumes for postoperative adjuvant radiotherapy in patients with stage C prostate cancer? Strahlenther Onkol. 2002 Mar;178(3):134-8. doi: 10.1007/s00066-002-0896-9. PMID 11962189
- [Background] Kotzerke J, Prang J, Neumaier B, Volkmer B, Guhlmann A, Kleinschmidt K, Hautmann R, Reske SN. Experience with carbon-11 choline positron emission tomography in prostate carcinoma. Eur J Nucl Med. 2000 Sep;27(9):1415-9. doi: 10.1007/s002590000309. PMID 11007527
- [Background] Pinto JT, Suffoletto BP, Berzin TM, Qiao CH, Lin S, Tong WP, May F, Mukherjee B, Heston WD. Prostate-specific membrane antigen: a novel folate hydrolase in human prostatic carcinoma cells. Clin Cancer Res. 1996 Sep;2(9):1445-51. PMID 9816319
- [Background] Smith-Jones PM, Vallabahajosula S, Goldsmith SJ, Navarro V, Hunter CJ, Bastidas D, Bander NH. In vitro characterization of radiolabeled monoclonal antibodies specific for the extracellular domain of prostate-specific membrane antigen. Cancer Res. 2000 Sep 15;60(18):5237-43. PMID 11016653
- [Background] Ghosh A, Heston WD. Tumor target prostate specific membrane antigen (PSMA) and its regulation in prostate cancer. J Cell Biochem. 2004 Feb 15;91(3):528-39. doi: 10.1002/jcb.10661. PMID 14755683
- [Background] Kinoshita Y, Kuratsukuri K, Landas S, Imaida K, Rovito PM Jr, Wang CY, Haas GP. Expression of prostate-specific membrane antigen in normal and malignant human tissues. World J Surg. 2006 Apr;30(4):628-36. doi: 10.1007/s00268-005-0544-5. PMID 16555021
- [Background] Milowsky MI, Nanus DM, Kostakoglu L, Sheehan CE, Vallabhajosula S, Goldsmith SJ, Ross JS, Bander NH. Vascular targeted therapy with anti-prostate-specific membrane antigen monoclonal antibody J591 in advanced solid tumors. J Clin Oncol. 2007 Feb 10;25(5):540-7. doi: 10.1200/JCO.2006.07.8097. PMID 17290063
- [Background] Hillier SM, Maresca KP, Femia FJ, Marquis JC, Foss CA, Nguyen N, Zimmerman CN, Barrett JA, Eckelman WC, Pomper MG, Joyal JL, Babich JW. Preclinical evaluation of novel glutamate-urea-lysine analogues that target prostate-specific membrane antigen as molecular imaging pharmaceuticals for prostate cancer. Cancer Res. 2009 Sep 1;69(17):6932-40. doi: 10.1158/0008-5472.CAN-09-1682. Epub 2009 Aug 25. PMID 19706750
- [Background] Olson WC, Heston WD, Rajasekaran AK. Clinical trials of cancer therapies targeting prostate-specific membrane antigen. Rev Recent Clin Trials. 2007 Sep;2(3):182-90. doi: 10.2174/157488707781662724. PMID 18474004
- [Background] Rajasekaran AK, Anilkumar G, Christiansen JJ. Is prostate-specific membrane antigen a multifunctional protein? Am J Physiol Cell Physiol. 2005 May;288(5):C975-81. doi: 10.1152/ajpcell.00506.2004. PMID 15840561
- [Background] Slovin SF. Targeting novel antigens for prostate cancer treatment: focus on prostate-specific membrane antigen. Expert Opin Ther Targets. 2005 Jun;9(3):561-70. doi: 10.1517/14728222.9.3.561. PMID 15948673